CLINICAL TRIAL: NCT00166803
Title: The Impact of Rosiglitazone on Regression of Atherosclerosis: A Serial 18F-Fluorodeoxyglucose Positron Emission Tomography Study
Brief Title: The Impact of Rosiglitazone on Regression of Atherosclerosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: no fund
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Pan-Chyr Yang, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 931110
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Mellitus, Atherosclerosis
Keywords: Diabetes Mellitus, PPARγ agonist, FDG PET
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone , 4 mg daily

SUMMARY:
Cardiovascular events are the leading cause of death in developed countries worldwide, including Taiwan. The disruption of atherosclerotic plaques and the subsequent formation of thrombi are currently recognized as the major cause of morbidity and mortality of cardiovascular diseases. Therefore, early detection of vulnerable plaques is clinically important for risk stratification and also to provide early treatment. Several imaging approaches have been adapted to detect vulnerable plaques, however, most of them are based on morphologic characteristics of atheroma. We hypothesize that PPARγ-induced plaque regression could be monitored clinically by use of 18FDG PET/CT approach, which could assess the inflammatory activity, and can be detected noninvasively earlier than previously reported.

DETAILED DESCRIPTION:
The early detection of vulnerable plaques is clinically important for risk stratification and also to provide early treatment.Inflammation is important in the both pathogenesis and outcome of atherosclerosis. Plaques containing numerous inflammatory cells, particular macrophages, have a high risk of rupture. Diabetes is a major risk factor for the development of atherosclerosis. The discovery of the peroxisome proliferator-activated receptor γ (PPARγ) gene led to the hope of favorably influencing the insulin resistance syndrome. The administration of PPARγ agonists have been shown to reduce insulin resistance, to reduce the expression of leptin, to lower plasma free fatty acid level and to lower blood pressure. Moreover, beyond the glucose effect, PPARγ agonists may theoretically affect atherosclerosis also through the inhibition of inflammatory cytokines secreted from the macrophage, such as IL-6, IL-1β, TNF-α, etc. These evidences highlight the possibility of PPARγ agonists could be have great impact on plaque regression.

18FDG is a glucose analogue that is taken up by cells in proportion to their metabolic activity. Several papers have reported the potential roles of metabolic imaging in the assessment of inflammatory vascular diseases, especially in large vessels. However, PET has limited spatial resolution. Recently, a combined PET/CT is emerged as a promising modality which could provide both anatomical and functional information. We hypothesize that PPARγ agonists-induced plaque regression could be monitored clinically by use of 18FDG PET/CT approach, and providing information of early efficacy PPARγ treatment caused by stabilization of vulnerable plaque without affecting the lumen size.

ELIGIBILITY:
Inclusion Criteria:

1. Type II DM patients who are aged 50 to 80 year-old with HbA1c between 7.0 to 10.0 %
2. Under ≤ 2 kinds of anti-diabetic drugs.

Exclusion Criteria:

1. Insulin use
2. Patients who receive any PPARγ agonist in recent one year.
3. Women of child-bearing potential are excluded (i.e. menopausal women or post-hysterectomy women are included in this study) due to radiation exposure in this study.
4. Significant concomitant disease such as active infection, malignancy, hepatic or renal dysfunction at the time of enrollment (i.e. T-Bil > 3 mg/dl，ALT > 2.5 times the upper limit of normal range and Creatinine > 3 mg/dl in our hospital).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Vulnerable plaque analyses by PET: Define plaque location and activity at baseline, and compare with the follow-up scans site by site. | 12 w

SECONDARY OUTCOMES:
1.Glycemic control after active treatment. (Fasting glucose level, HbA1c) | 12 w
2.Biomarkers:hs-CRP, MMP-1, MCP-1. | 12 w

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Shiung Yang, MD, phD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan